CLINICAL TRIAL: NCT04211688
Title: Real-world Effectiveness of a Combined Group-individual Schema Therapy for Borderline Personality Disorder: A Pragmatic Randomized Clinical Trial
Brief Title: Effectiveness of a Combined Group-individual Schema Therapy for Borderline Personality Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari del Maresme (Other)
Collaborators: Department of Health, Generalitat de Catalunya (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 32/16
Record Dates: First submitted 2019-12-19; First posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Borderline Personality Disorder; Randomized Controlled Trial
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined individual + group Schema therapy (Experimental): Those who will receive both individual plus group schema therapy
  Interventions: Behavioral: Group Schema therapy; Behavioral: Individual Schema therapy
- Only group Schema therapy (Active Comparator): Those who will receive group schema therapy
  Interventions: Behavioral: Group Schema therapy

INTERVENTIONS:
Behavioral: Group Schema therapy — Bimonthly outpatient psychotherapy delivered in individual setting
Behavioral: Individual Schema therapy — weekly outpatient psychotherapy delivered in group setting
  Arms: Combined individual + group Schema therapy

SUMMARY:
Background and Objectives: Schema therapy has been shown to be of benefit in treating borderline personality disorder. However, it is still unclear what the most suitable treatment implementation format is and to what extent therapeutic gains may be generalizable to regular healthcare settings with limited resources.

Methods: A pragmatic randomized controlled trial was conducted ona representative Spanish sample of outpatients with a DSM-5 main diagnosis of borderline personality disorder. Patients were allocated either to a combined (group plus individual) schema therapy format (n=40) or to a group-only schema therapy format (n=40). Borderline personality disorder severity was the primary outcome, with other clinical variables considered as secondary outcomes (e.g., early maladaptive schemas, functioning). The assessment protocol included baseline, post-treatment (after 12months of treatment), and six-month follow-up evaluations. Data was analyzed through a two-way repeated measures ANOVA. Limitations were a limited follow-up assessment and the absence of multi-center data that detracted from the long-term stability and generalizability of the findings.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 criteria for borderline personality disorder
* Aged 18 to 65 years

Exclusion Criteria:

* Psychotic disorders (except short, reactive psychotic episodes)
* Bipolar disorder (current hypo-manic or mixed episode)
* Antisocial personality disorder
* Substance intoxication
* Mental retardation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
BPD (borderline personality disorder) symptomatology | 18 months
  Severity of borderline symptomatology as measured by a single score from the BSL-23 scale (range: 0-92; the higher the score, the more severe the BPD severity).

SECONDARY OUTCOMES:
global functioning | 18 months
  Severity of dysfunction as measured by a single score from the WHOQoL scale (range: 0-100; the higher the score, the more severe the global dysfunction).
early maladaptive schemas | 18 months
  Severity of maladaptive schemas as measured by a single score from the YSQ scale (range: 0-450; the higher the score, the more severe the EMS severity).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zanarini MC. Psychotherapy of borderline personality disorder. Acta Psychiatr Scand. 2009 Nov;120(5):373-7. doi: 10.1111/j.1600-0447.2009.01448.x. PMID 19807718
- [Result] Farrell, J. M., & Shaw, I. A. (2012). Group schema therapy for borderline personality disorder. A step-by-step treatment manual with patient workbook. West Sussex, UK: Wiley-Blackwell.